CLINICAL TRIAL: NCT04462757
Title: Subcutaneous and Intravenous IL-1Ra (Anakinra) in COVID-19 Infection - Feasibility & Pharmacokinetics/Pharmacodynamics Study
Brief Title: SCIL-1Ra in COVID-19 Feasibility & PK/PD
Acronym: SCIL_COV19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patients in the trial population from which to recruit and lack of funding
Sponsor: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 282110; 2020-001636-95 (EudraCT Number)
Record Dates: First submitted 2020-06-12; First posted 2020-07-08 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of two arms:-
  * Subcutaneous arm: 100mg anakinra SC will be administered subcutaneously at consistent times that are convenient and practical for the patients and research/nursing staff providing there is a minimum 8 hours and maximum 16 hours between administrations.
  * Intravenous arm: 100mg anakinra in 100mL 0.9% NaCl will be administered intravenously four times a day every 6 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcutaneous Arm (Active Comparator): 100mg anakinra SC will be administered subcutaneously at consistent times that are convenient and practical for the patients and research/nursing staff providing there is a minimum 8 hours and maximum 16 hours between administrations.
  Interventions: Drug: Anakinra 100Mg/0.67Ml Inj Syringe
- Intravenous Arm (Active Comparator): 100mg anakinra in 100mL 0.9% NaCl will be administered intravenously four times a day every 6 hours.
  Interventions: Drug: Anakinra 100Mg/0.67Ml Inj Syringe

INTERVENTIONS:
Drug: Anakinra 100Mg/0.67Ml Inj Syringe — 100 mg interleukin-1 receptor antagonist (r-meth-Hu-IL-1Ra), anakinra; marketed as Kineret® in 0.67 mL prefilled syringe for single use
  Other Names: Kineret

SUMMARY:
The current COVID-19 pandemic is a worldwide healthcare crisis. Of concern is the large number of patients that are/will require mechanical ventilation, and the associated strain that this will place on healthcare resources. At present, there are no specific therapeutic interventions directed at COVID-19 infection. However, observational data suggest that there is a subgroup of patients that demonstrate a hyperinflammatory response in response to COVID-19 and have a higher requirement for Critical Care and higher mortality.

There is a strong case for the use of the naturally occurring anti-inflammatory cytokine interleukin-1 receptor antagonist (IL-1Ra) in these patients. Anakinra is a recombinant form of IL-1Ra that is licensed for clinical use. Success of use of anakinra in COVID-19 trials will be greatly enhanced by robust scientific evidence and established pharmacokinetics which inform the most effective dosing regimens. The latter is especially important when, as in the case of anakinra, drug supplies are limited, the drug has short half-life and clinical ease of application is critical.

DETAILED DESCRIPTION:
The investigators plan a small trial of an existing drug in patients with COVID-19 at Salford Royal NHS Foundation Trust (SRFT) and Manchester Foundation Trust (MFT). The investigators will recruit patients with suspected or confirmed COVID-19 infection within 24 hours of being transfer in a Critical Care department. The investigators have been testing interleukin-1 receptor antagonist: IL-1Ra (known as Anakinra) for many years. Marketed as a treatment for rheumatoid arthritis and for some rare autoimmune diseases, we have shown Anakinra also reduces or blocks inflammation in a number of other conditions e.g. stroke and brain haemorrhage. The investigators have found it to be safe, easily administered and well tolerated. As part of the global response to the SARS-COV-2 pandemic, researchers have identified drugs that repurposing existing drugs. Anakinra has been proposed as a candidate therapy for COVID-19 and will be used in REMAP-CAP clinical trial as an intravenous (IV) therapy four times daily (qds). Whilst there is uncertainty about the therapeutic benefits, the investigators wish to explore the theory that they can achieve comparable concentrations in the blood using a subcutaneous (SC) injection twice daily (bd), as observed with IV therapy qds. We will randomise up to 40 patients to receive either SC Anakinra twice daily or IV Anakinra four-times daily for 14 days (or until discharge from CCU). They will measure changes in biomarkers in both groups and use the data to inform a mathematical model to simulate the effect the drug may have on the body. The aim is to the provide evidence that a lower dose SC Anakinra is as effective as higher dose IV.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 or above.
* Clinically suspected/proven COVID-19.
* Requiring organ support with one or more of:
* Non-invasive or invasive ventilatory support
* Receiving infusion of vasopressor or inotropes or both.
* No concomitant health problems that, in the opinion of the PI or designee in agreement with the treating clinician, would interfere with participation, administration of study drug or assessment of outcomes including safety.

Exclusion Criteria:

* More than 24h has elapsed since CCU admission.
* Death is deemed to be imminent and inevitable during the next 24h.
* One or more of: the patient, substitute decision-maker or the attending physician are not committed to full active treatment.
* Known condition resulting in ongoing immunosuppression including neutropenia (count < 1.5 x 10^9/L) prior to hospitalisation, malignancy, latent tuberculosis or chronic liver disease (if known).
* Previous or current treatment with anakinra or medication suspected of interacting with anakinra, listed in the drug SmPC, known at the time of trial entry or previous participation in this trial.
* Known to have received active treatment in a clinical trial of an investigational immunomodulatory agent (not including corticosteroids) within 30 days prior to study entry.
* Known to be pregnant or breast feeding or inability to reliably confirm that the patient is not pregnant.
* Known allergy to anakinra or any of the excipients listed in the drug SmPC
* Known allergy to other products that are produced by DNA technology using the micro-organism E. coli (e.g. Escherichia coli derived protein).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Plasma IL-1Ra levels | 1 week
  Plasma IL-1Ra levels from Day 1 to Day 7 following administration of SC anakinra in patients with SARS-CoV-2
Plasma IL-6 levels | 1 week
  Plasma IL-6 levels from Day 1 to Day 7 following administration of SC anakinra in patients with SARS-CoV-2

SECONDARY OUTCOMES:
Plasma markers | 2 weeks
  Plasma markers including IL-6 from Day 1 to Day 14 in all participants
Plasma markers | 2 weeks
  Plasma markers including CRP from Day 1 to Day 14 in all participants
Plasma markers | 2 weeks
  Plasma markers including CXCL9 from Day 1 to Day 14 in all participants
Plasma markers | 2 weeks
  Plasma markers including IL-1 from Day 1 to Day 14 in all participants
Plasma markers | 2 weeks
  Plasma markers including IL-2 from Day 1 to Day 14 in all participants
Plasma markers | 2 weeks
  Plasma markers including HMBG-1 from Day 1 to Day 14 in all participants
Plasma markers | 2 weeks
  Plasma markers including IL-33 from Day 1 to Day 14 in all participants
Safety Endpoints related to the Serious adverse reactions of the IMP | 2 weeks
  Safety endpoints include:
  a. Severe fatal or life-threatening serious adverse reactions (duration of IMP plus 30h from last dose).
Safety Endpoints related to the anaphylactic reactions of the IMP | 2 weeks
  Safety endpoints include:
  b. Anaphylactic/anaphylactoid reactions (duration of IMP plus 30h from last dose).
Safety Endpoints related to neutropenia caused by the IMP | 2 weeks
  Safety endpoints include:
  c. Severe neutropenia (< 1.5 x 109 /L) (duration of IMP)
Safety Endpoints related to any severe laboratory abnormalities | 2 weeks
  Safety endpoints include:
  d. IMP related severe laboratory abnormalities (duration of IMP)
Feasibility endpoints related to IMP and deviations | 2 weeks
  Feasibility endpoints include protocol deviations in terms of timing and delivery of scheduled medication.
Exploratory Data on Clinical efficacy by time to recovery | 4 weeks
  Exploratory data on clinical efficacy as defined by:
  a. Time to recovery defined by hospital discharge or improvement of two points on the ordinal scale: not hospitalised; hospitalised without need for supplemental oxygen; requiring supplemental oxygen; requiring HFNC or non-invasive mechanical ventilation; requiring ECMO or mechanical intervention; dead. Improvement mechanical ventilation (from recruitment to time of ventilation)
Exploratory Data on Clinical efficacy | 4 weeks
  Exploratory data on clinical efficacy as defined by:
  b. Ventilation free days (at 28 days)
Exploratory Data on Clinical efficacy of the ordinal scale | 4 weeks
  Exploratory data on clinical efficacy as defined by:
  c. Status on the above ordinal scale (at 14 and 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Felton, Dr, Principal Investigator — University of Manchester
Locations (2):
- United Kingdom (2):
  - Manchester Univesity NHS Foundation Trust, Manchester
  - Salford Royal NHS Foundation Tust, Salford

IPD SHARING:
Plan to Share IPD: No